CLINICAL TRIAL: NCT06721819
Title: The SCOPE Trial: Sleep, Cognition, and Pain Bundle Vs. ERAS-cardiac for Postoperative Delirium
Acronym: SCOPE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Massachusetts General Hospital (Other); Ohio State University (Other); Columbia University (Other)
Responsible Party: Principal Investigator, Balachundhar Subramaniam, Professor of Anaesthesia, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DE-2023C1-31327
Record Dates: First submitted 2024-11-25; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Delirium, Postoperative; Delirium in Old Age
Keywords: Delirium; PostOperative; Cardiac Surgery
MeSH Terms: conditions — Emergence Delirium; Delirium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sleep Hygiene, brain games, and IV Acetaminophen bundle intervention (Experimental): Preoperative Intervention: Two weeks of following a sleep hygiene protocol and 10 hours minimum of playing brain games.
  Cognitive Exercise: Patients will be given an iPad, which will be pre-installed with access to Lumosity, a cognitive exercise software application. Participants will be instructed to try and complete 1 hour of Lumosity exercise daily prior to surgery, with a pre-operative cognitive exercise goal of 10 hours.
  Sleep Hygiene: Preoperatively, investigators will deliver the digital CBT-I, (Cognitive Behavioral Therapy- Insomnia) over 2 weeks before surgery and in parallel to cognitive exercise.
  Postoperative Intervention: Eight doses of IV acetaminophen at 1000g each dose delivered every 6 hours for the first 48 hours within 1 hour of admission to CVICU. Acetaminophen administration in any form other than the blinded study medication during this time will not be allowed.
  Interventions: Combination Product: Sleep Hygiene, Brain Game, and IV Acetaminophen Intervention
- ERAS Protocol with three doses IV Acetaminophen (Active Comparator): No preoperative intervention and three doses of IV acetaminophen (as following ERAS protocol) at 1000mg per dose within 48 hours post operatively. Control patients will be on intravenous acetaminophen for the first 24 hours (three doses at 8 hourly intervals).
  Interventions: Drug: Control

INTERVENTIONS:
Combination Product: Sleep Hygiene, Brain Game, and IV Acetaminophen Intervention — Preoperative Sleep Hygiene and Brain game followed by post operative IV acetaminophen administration
  Other Names: CBT-I; Lumosity; IV-Acetaminophen
  Arms: Sleep Hygiene, brain games, and IV Acetaminophen bundle intervention
Drug: Control — Three doses of IV acetaminophen (as following ERAS protocol) at 1000mg per dose within 48 hours post operatively.
  Arms: ERAS Protocol with three doses IV Acetaminophen

SUMMARY:
Sleep disturbances, cognitive reserve, and continuing pain and inflammation are other risk factors contributing to delirium (confusion and agitation) and neurocognitive decline (in the long term) following heart surgery. Investigators aim to test a bundle of sleep optimization, cognitive exercise before surgery, and extended pain relief for 48 hours with intravenous acetaminophen combined with enhanced recovery after surgery protocols (SCOPE bundle). SCOPE will fill significant gaps in evidence by testing the value of a patient and care-provider-focused intervention that can potentially minimize POD and improve outcomes (cognitive & physical function, sleep quality, pain, depression or anxiety, and survival) important to patients and families.

The SCOPE trial will address many heart surgery outcome-related questions commonly asked by patients:

What can I do to reduce my chances of developing confusion, hallucinations, or delirium after surgery? How can I best prepare before surgery to improve my long-term health and avoid disability? Are there exercises I can participate in that improve my sleep, pain, and mood after surgery? Intellectual pursuits, physical activity, and social interactions support cognitive reserve, while poor health, poor sleep hygiene, poor nutrition, and mental health disease can diminish reserve. Various interventions with different intensities and timing to augment cognitive reserve have been associated with positive outcomes on neuropsychological testing. Adaptive video gaming for as little as 10 hours leads to the maintenance of independence in activities of daily living and sustained improvements in speed of processing, attention, and working memory in older people. Likely through the increased cognitive reserve, perioperative brain exercise aims to protect against morbid cognitive recovery after surgery.

Sleep is vital for memory and cognitive function. Poor sleep traits in older adults that are potentially modifiable, including short/long duration, daytime napping, and associated sleepiness, led to an almost 2-fold increase in delirium risk. Patients will complete an evidence-based course on healthy sleep habits and will complete guided exercises designed to restructure behaviors and thinking. They are encouraged to follow a set of recommendations to improve their sleep (e.g., optimal sleep duration, advice for habits such as daytime napping, maintaining a regular sleep schedule, avoiding caffeine, regular daylight exposure, dimming lights or electronics and relaxation and thought exercises for optimal sleep); many of these sleep behaviors have been strongly linked to increased risk for cognitive decline. Investigators propose that sleep optimization before AND after (an established best practice sleep bundle) surgical insult will contribute to cognitive reserve leading to decreased delirium risk and key patient-centered outcomes (postoperative sleep, pain, cognition, mood, and survival).

Inadequate pain relief and opioids are both risk factors for delirium. Surgery on the chest is a significant pain source. Approximately 30-75% of patients suffer from moderate to severe pain in the postoperative period. Almost half of the patients have severe pain at rest, and three-quarters have severe pain during coughing and movement. Pain and inflammation are closely biochemically linked.

Sleep, brain exercise, and adequate pain control with opioid-sparing can be additive or synergistic interventions to prevent delirium following heart surgery.

Investigators propose three specific aims by conducting a 1:1 randomized controlled trial in 406 heart surgery patients 60 or older undergoing heart surgery. They will be administered perioperative sleep optimization, brain exercise training, and intravenous acetaminophen over 48 hours. A trained expert will administer the sleep and cognitive exercise protocols at least two weeks before surgery. This expert will handhold the patients for two weeks until the surgery. Thus, the gains made before surgery with better sleep quality and improved brain reserve will be sustained with postoperative pain control to lower the ongoing inflammation. Through this trial, investigators will evaluate if the SCOPE bundle can reduce 1) in-hospital delirium, 2) long-term (one, six, and twelve months) cognitive, physical, and self-care function, and 3) barriers to implementation of this bundle.

Currently, no options are routinely available to patients to optimize their sleep and cognition before cardiac surgery. The proposed research is significant because it will be the first to test the bundled behavioral intervention approach (sleep optimization, brain exercise) before surgery with extended, scheduled pain management with non-opioids following surgery. The SCOPE trial will yield relevant and immediately actionable data to improve care for over 900,000 adults in the U.S. each year.

DETAILED DESCRIPTION:
Background and Significance: Cardiac surgery is performed on more than 900,000 adults in the U.S. each year, with significant cognitive consequences for individuals and society. Postoperative delirium (POD) is a common and costly complication after cardiac surgery. POD prevention is a priority for patients, families, and clinicians. Cognitive reserve is a significant contributor to POD risk. Despite many successes of Enhanced Recovery After Surgery (ERAS) initiatives to improve patient outcomes, incorporating cognitive-protective strategies into protocols remains limited by lack of evidence. The SCOPE Trial (Sleep, Cognition, and Pain bundle vs. ERAS-cardiac (enhanced recovery after cardiac surgery) for POD) will fill significant gaps in delirium prevention evidence by testing the value of a patient and care-provider-focused intervention that can potentially minimize POD. Study Aims: Investigators hypothesize that the intervention bundle (multicomponent combination of non-pharmacological (pre- and post-operative sleep optimization and cognitive exercise) and pharmacological (extended postoperative opiate-sparing pain control with intravenous (IV) acetaminophen for 48 hours) will decrease POD incidence and improve outcomes compared to standard ERAS protocols alone. Investigators hypothesize that the bundle increases 1) resistance to circadian disruption, 2) improved neuronal function, and 3) cognitive reserve. Investigators will determine differences in incidence, duration, and severity of POD (Specific Aim 1) and postoperative functional status, cognition, sleep, pain, and mood between study groups 1, 6, and 12 months following cardiac surgery (Specific Aim 2). Investigators will evaluate implementation barriers for our multicomponent SCOPE bundle and acceptability and feasibility (Specific Aim 3). Study Description: The SCOPE trial is a multicenter randomized, multi-component, superiority trial in older patients (at least 60 years) undergoing non-emergent coronary artery bypass grafting with or without valves or isolated valve surgery with 1:1 allocation using permuted block randomization of variable block sizes 2, 4, and 6 (406 patients equally divided at four tertiary care centers across the U.S (Beth Israel Deaconess Medical Center (n=106), Massachusetts General Hospital (n=100), Columbia University (n=100) and Ohio State University Medical Center (n=100). Patients with alcohol abuse, hypersensitivity to acetaminophen, and severely depressed left ventricular ejection fraction (<30%) will be excluded. Enrolled participants will receive either the SCOPE regimen at least 2 weeks before surgery and scheduled postoperative acetaminophen analgesia for the first 48 hours (plus ERAS)) or the standard-of-care ERAS regimen only.

1. Investigators will use a shorter form of our existing clinical CBT program for insomnia (4 hybrid sessions), delivered over two weeks before cardiac surgery to optimize sleep. Investigators will also check in with patients to establish sleep preferences during postoperative recovery, e.g., usual sleep schedule, noise reduction aids, temperature, light, and music preferences. Key components that can be effectively taught and implemented quickly based on our clinical experience include, stimulus control, relaxation techniques, sleep hygiene education, and cognitive restructuring to address sleep-related anxiety misconceptions and relaxation techniques. The Control group will be given a sleep hygiene education tip sheet only.
2. To optimize cognitive function, intervention patients will be asked to complete 10 hours of preoperative tablet-based brain exercise using gaming software focused on memory, speed, attention, flexibility, and problem-solving. This has been designed and integrated with the above sleep intervention to streamline patient experience and decrease burden and maximize retention. A prehabilitation specialist will deliver these interventions.
3. SCOPE-bundle patients will receive eight doses of IV acetaminophen over 48 hours (compared to standard pain management for ERAS includes three doses of IV acetaminophen over 24 hours).

The primary study outcome is POD incidence within seven days or until discharge following cardiac surgery, whichever occurs first, as determined by the Confusion Assessment Method (CAM) or CAM-ICU, supplemented with charted delirium. Secondary outcomes include POD duration (number of days), severity (CAM-Severity), length of postoperative stay (days), and mortality (30 days). Additional secondary outcomes assessed up to 12 months post-surgery include (pain (analgesia requirements, Verbal Rating Pain Scale), mood (Geriatric Depression Scale), functional recovery (Instrumental Activities of Daily Living and Medical Outcomes Study Short Form 12), and sleep quality (Pittsburgh Sleep Quality Index and objective metrics via sleep diary, and actigraphy). Secondary outcomes of determinants of bundle implementation, feasibility, and acceptability of implementation will be evaluated within the integrated Promoting Action on Research Implementation in Health Services (i-PARIHS) framework at the start and conclusion of the study

ELIGIBILITY:
Inclusion Criteria:

* Planned cardiac surgery [CABG with or without valve, isolated valve surgery] requiring median sternotomy and full CPB at least two weeks in the future.

  * 60 years of age.

Willingness to use a provided tablet and wearable devices and commit at least 1 hour amount of time per day before surgery to complete interventions (psCBT/cognitive activity/exercise) if randomized to experimental group.

Exclusion Criteria:

* Pre-operative left ventricular ejection fraction (LVEF) < than 30%

Emergent procedures

Isolated aortic surgery

Liver dysfunction (ALT or AST > 4 times the upper limit of local normal; all patients will have a baseline liver function test information or history and exam suggestive of jaundice or both)

Known hypersensitivity to the study drugs

Active (in the past year) history of alcohol abuse (≥ 5 drinks/day for men or ≥ 4 drinks/day for women) Any history of alcohol withdrawal or delirium tremens

Delirium at baseline

English language Limitations

Physician refusal

Chronic opioid use for chronic pain conditions with tolerance (total dose of an opioid at or more than 30 mg morphine equivalent for more than one month within the past year)

Significant visual impairment

Prisoner

Severe OSA in the past year (AHI is greater than 30 (more than 30 episodes per hour)) or ESS of 18 or more

Co-enrollment with non-approved interventional trial

Severe cognitive impairment (MOCA < 10) or medications for cognitive decline

Recent treatment for insomnia with CBT-I within the last 6 months

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2029-06-30 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Delirium Incidence | Seven days following cardiac surgery or until discharge of patient from the hospital. This can be anywhere from 3-7 days post operatively
  Positive CAM (Confusion Assessment Method) evaluation. : The Confusion Assessment Method (CAM) is a standardized evidence-based tool that enables non-psychiatrically trained clinicians to identify and recognize delirium quickly and accurately in both clinical and research settings. The CAM includes four features found to have the greatest ability to distinguish delirium from other types of cognitive impairment. Each feature is scored as present or absent. Delirium is considered present based on the CAM diagnostic algorithm: presence of (acute onset or fluctuating course -AND- inattention) -AND EITHER- (disorganized thinking or altered level of consciousness)

SECONDARY OUTCOMES:
Severity of Delirium | Seven days following cardiac surgery or until discharge of patient from the hospital. This can be anywhere from 3-7 days post operatively
  CAM- S (Confusion Assessment Method- Severity) score. A delirium severity rating scale based on the additive scoring of symptoms rated in the CAM long form (Confusion Assessment Method). The CAM-S is intended to be used in addition to the original CAM algorithm. The scale for CAM-S is from 0-19 with 0 being the least severe and 19 being the most severe.
Duration of Delirium | Seven days following cardiac surgery or until discharge of patient from the hospital. This can be anywhere from 3-7 days post operatively
  The total number of days patient is CAM (Confusion Assessment Method) positive following cardiac surgery

OTHER OUTCOMES:
Incidence of delirium in patients with active alcohol and drug abuse | Seven days following cardiac surgery or until discharge of patient from the hospital. This can be anywhere from 3-7 days post operatively
  Confusion Assessment Method (CAM) positive result in patients who have a history of active alcohol and drug abuse
Incidence of delirium in patients with preoperative neurocognitive impairment, Parkinson's and Alzheimer's disease Incidence of delirium in patients with preoperative neurocognitive impairment, Parkinson's and Alzheimer's disease | Seven days following cardiac surgery or until discharge of patient from the hospital. This can be anywhere from 3-7 days post operatively
  Confusion Assessment Method (CAM) positive result in patients who have a medical history with preoperative neurocognitive impairment, and/or Parkinson's disease, and/or Alzheimer's disease
Intraoperative hypotension | Seven days following cardiac surgery or until discharge of patient from the hospital. This can be anywhere from 3-7 days post operatively
  Investigators will explore if during the surgery the patient has any hypotension (systolic blood pressure below 90 and diastolic blood pressure 60), it has an effect on postoperative delirium incidence
Functional status | Enrollment in trial to 12 months post discharge from hospital
  Participants functional status is assessed by IADL and SF-12. The Lawton Instrumental Activities of Daily Living Scale (IADL) is an appropriate instrument to assess independent living skills. The instrument is most useful for identifying how a person is functioning at the present time, and to identify improvement or deterioration over time. Clients are scored according to their highest level of functioning in that category. A summary score ranges from 0 (low function, dependent) to 8 (high function, independent) for women, and 0 through 5 for men. The Short Form Health Survey (SF-12) is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.
Pain scores | Participant is admitted to the Intensive Care Unit post cardiac surgery until 12 months post hospital discharge.
  Assessment of pain while subject is enrolled in trial using VPRS (verbal pain rating scale). The Numerical Rating Pain Scale is a simple pain scale that grades pain levels from 0 (No pain), 1,2, and 3 (Mild), 4,5, and 6 (Moderate), 7,8, and 9 (Severe) to 10 (Worst Pain Possible).
Length of stay and mortality | Once the patient is admitted into the intensive care unit (ICU) post surgery until they are discharged from the hospital. This can be anywhere from 1-30 days post operatively.
  The length of stay will be calculated by the number of days the patient is in hospital post surgery till discharge. The mortality will be recorded if the participant passes away during their in hospital stay.
Assessment of feasibility of implementation of intervention | Before the study is initiated and end of data collection for the study
  To see if implementation of intervention bundle will be feasible in clinical care settings using the Integrated-Promoting Action on Research Implementation in Health Services (I-PARIHS) framework. This framework will guide evaluation and interpretation of determinants (facilitators and barriers) of our bundles' implementation. To elucidate facilitators and barriers within each domain, additional qualitative data will be gathered via semi-structured individual interviews and focus groups of participants/caregivers and clinicians from each site before study initiation and at the end of the study.
Sleep Quality | From time of enrollment to 12 months post discharge from hospital
  Sleep quality is measured by PSQI, ESS, and ISI. The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. Scores for each question range from 0 to 3, with higher scores indicating more acute sleep disturbances. The Epworth Sleepiness Scale (ESS) is a self-administered questionnaire with 8 questions. The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life (ASP). Insomnia Severity Index (ISI) is designed as a brief screening tool for insomnia, the seven-item questionnaire asks respondents to rate the nature and symptoms of their sleep problems using a Likert-type scale. Responses can range from 0 to 4, where higher scores indicate more acute symptoms of insomnia.
Mood and Stress | From time of enrollment to 12 months post discharge from hospital
  Investigators will use Geriatric Depression Scale (GDS) for mood assessment and Post-Traumatic Stress Disorder Checklist for DSM-5 (PCL-5) to assess stress. A Short Form GDS consisting of 15 questions. Of the 15 items, 10 indicated the presence of depression when answered positively, while the rest (question numbers 1, 5, 7, 11, 13) indicated depression when answered negatively. Scores of 0-4 are considered normal, depending on age, education, and complaints; 5-8 indicate mild depression; 9-11 indicate moderate depression; and 12-15 indicate severe depression. The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. Items are summed to provide a total severity score (range 0-80) with a cutoff score between 31-33 can be used for a provisional PTSD diagnosis.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Columbia University Irving Medical Center, New York, New York
  - The Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No